CLINICAL TRIAL: NCT01416168
Title: Pilot Study of a Geriatric Intervention After Colorectal and Lung Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Tampa General Hospital (Other); University of South Florida (Other); Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-15641
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
Keywords: Colon; Geriatric; McCorkle Model; Questionnaire
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Arm (No Intervention): Usual post-surgical care
- Intervention arm (Experimental): In addition to usual post-surgical care, the patients will receive a 4 week geriatric nurse practitioner-centered intervention, based on the McCorkle model.
  Interventions: Other: McCorkle Model Intervention

INTERVENTIONS:
Other: McCorkle Model Intervention — The intervention will consist each week in a home visit and a phone call. The GNP conducting the home visit will identify current problems using a comprehensive geriatric assessment (CGA) and record problems on the Intervention and Recommendation Data Sheet. In addition, the cases will be reviewed at a weekly Intervention Team meeting between the intervention GNP (VM, CV), the geriatrician (VP), and the intervention PI (JO). That team meeting will also record how intervention goals for the various problems are met, using the instruments and criteria developed during our pilot study5. To ensure optimal consistency and an up-to-date evidence-based approach over the 4 years of the intervention, treatment recommendations will be offered according to national evidence-based treatment guidelines.
  Arms: Intervention arm

SUMMARY:
Surgery for colorectal cancer is a major surgery. People above the age of 60 tend to have a higher risk of complications. Some studies indicate that senior cancer patients might benefit from a home support after surgery by a geriatric nurse practitioner and a team, beside their usual post-operative care. The investigators team is planning a large study to assess whether this approach could help patients with colorectal cancer recover better from their surgery, get better cancer treatment after that (e.g. chemotherapy), and possibly live longer. This study you are asked to take part in is a pilot for this large study.

DETAILED DESCRIPTION:
Our key background data come from the randomized study conducted by McCorkle et al.

After evaluation testing, patients will be randomly assigned (similarly to a coin toss) to one of two possible follow-up groups. One would be a regular post-surgery care group (control group), the other will have in addition a support by geriatric nurse practitioner (intervention group).

Patients who are assigned to the intervention group: once they arrive home, in addition to their normal post-surgery care, will receive a once a week home visit by a geriatric nurse practitioner (GNP). The GNP will also call the patient once a week in between. The GNP will check any problem patients may have during their recovery and provide or organize care for it. The GNP has a checklist of problems to address so that we can reliably reproduce our intervention in other patients. The GNP will work together with the patient's various doctors and caregivers, as well as a geriatric team. Some of the visits or the telephone calls maybe tape-recorded so that the research team can evaluate the information provided to the patient. We will record any complication patients might have from surgery.

No matter which treatment group the patient is assigned to, at the end of a 4 weeks period, we will repeat the tests we did at the beginning to see how they change.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer, stage III or IV, confirmed by histology
* Abdominal surgery by a University of South Florida (USF) surgeon at Moffitt Cancer Center or Tampa General Hospital (TGH)
* Age 60 years and older
* Informed consent
* Living within a one (1) hour radius of Moffitt

Exclusion Criteria:

* Discharge planned to a rehabilitation facility or a nursing home
* Unable to answer the questionnaires (e.g. because of cognitive impairment, blindness, deafness)
* Post-operative inpatient stay >one (1) month

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | 30 days per participant
  The primary end-point for the pilot will be the feasibility of the intervention, measured as follows:
  * A compliance of >=90% with the intervention table on page 17
  * A success rate (improvement or resolution of problems) of >= 80%
  * A completion rate of >=90% of the initial and final study questionnaires

SECONDARY OUTCOMES:
Whether the Intervention is Faithful to Dr. McCorkle's Original Intervention | 30 days per participant
  Aim 2 will be judged qualitatively. Dr. Ruth McCorkle and Dr. Janine Overcash will judge whether the intervention is faithful enough to Dr McCorkle's original intervention and whether it can be carried effectively by the trained personnel.
A Successful Collection and Testing of >=90% of the Samples Tested | 30 days per participant
  Aim 3 will be judged by assessing the percentage of tests that could or not be performed on the Moffitt patients.
Effect Size Estimates for Within-group Changes Between Baseline and 1-month | 30 days per participant
  Aim 4 will be assessed by the activities of daily living (ADL), instrumental activities of daily living (IADL), complications and FACT-colorectal (FACT-C) v.4 questionnaires at baseline and end of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Extermann, M.D., Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States